CLINICAL TRIAL: NCT06739863
Title: Evaluation of Different Healthcare Waste Management Practices and Problems Among Primary and Secondary Hospitals in Mianwali
Brief Title: Evaluation of Healthcare Waste Management Practices and Problems Among Primary and Secondary Hospitals
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Fall22/001
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthcare Associated Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Desc
  Interventions: Other: healthcare waste management

INTERVENTIONS:
Other: healthcare waste management — To evaluate and compare the healthcare waste management practices in primary and secondary hospital Mianwali.
  Focuses on assessing the current methods of waste disposal, segregation, treatment, and overall management in healthcare settings at two different levels of care: primary and secondary hospitals.

SUMMARY:
Healthcare waste is defined as the total waste stream from a healthcare facility. Most of it (75-90%) is similar waste to domestic waste and is known as healthcare general waste and is made up of paper, plastic packaging, food preparation etc. But as a similar proportion (10-25%) is hazards waste and requires special treatment. If these two categories of wastes are not separated properly then the entire volume of healthcare waste is considered as infectious and hazardous to human health and can result in disease and injury so it is necessary to set up a safe and integrated management system.

In this cross-sectional study public hospitals of Mianwali City will be selected by simple random sampling for observation of practices of hospital waste management.

DETAILED DESCRIPTION:
The data will be collected through structured Questionnaire and possibly on-sit Quantitative data on waste management practices, types of waste, compliance with regulations, and perceived challenges.

ELIGIBILITY:
Inclusion Criteria:

* Operation theatre Staff
* intensive care staff and labour room staff and laboratory room staff will be included.
* Doctors, Nurses, Nursing assistants, OT Technician, Maid's helpers, and sanitary workers.

Exclusion Criteria:

* Management staff will be excluded.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: included heathcare workers in hospitals including Operation theatre Staff, intensive care staff and labour room staff and laboratory room staff will be included, Doctors, Nurses, Nursing assistants, OT Technician, Maid's helpers, and sanitary workers
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
T.Test | 12 Months
  This is the test statistic that help us how far apart the means of the two groups are, in terms of the standard error of the difference between them. A larger t-value indicates a larger difference between the groups relative to the variation within the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- all Shumali Tehsil piplan District Mianwali, Mianwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No